CLINICAL TRIAL: NCT05784038
Title: Observational, Prospective, Cohort Study of Mpox Infection in Brazil - NETPOX Cohort
Brief Title: Observational, Prospective, Cohort Study of Mpox Infection in Brazil (NETPOX)
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: NETPOX
Record Dates: First submitted 2023-03-07; First posted 2023-03-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Monkeypox; MPOX
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples With DNA — Blood samples; Urine; oropharynx and Skin Lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human cases of monkeypox confirmed by PCR: Laboratory-confirmed mpox infection is defined as determined by polymerase chain reaction assay (PCR), culture, or antigen test obtained from a sample collected from blood, oropharynx, anal or skin lesion within 5 days of inclusion.
  Interventions: Diagnostic Test: Viral genomic; Diagnostic Test: Untargeted Metabolomics

INTERVENTIONS:
Diagnostic Test: Viral genomic — Evaluation of mpox viral genomic
Diagnostic Test: Untargeted Metabolomics — Evaluation of metabolomics of the total plasma, oropharynx, and skin samples.

SUMMARY:
The study is a prospective cohort that evaluates the clinical and immune-metabolic variables that may be linked to the risk and severity of the infection or even hospitalization or death in patients infected with the Mpox virus in Brazil. The expectation is to include at least 80 patients over six months, with a follow-up of 90 days from inclusion, through contact via decentralized visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years with confirmed MPOX infection.

(laboratory-confirmed monkeypox infection is defined as determined by PCR, culture, or antigen test obtained from a sample collected from blood, oropharynx, anal or skin lesion within 4 days of randomization)

Exclusion Criteria:

* Inability to provide informed consent;
* Patient who, judging by the study team, does not have a condition for decentralized follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Individuals who have risk factors for mpox infection in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composed of incidence of rash, fever, adenopathy, general pain, chills, weakness, occurrence of hospitalization, and neurological repercussions | Up to 90 days after the inclusion
  symptoms' incidence in participants with mpox infection

SECONDARY OUTCOMES:
Death | Up to 90 days after the inclusion
  Incidence of death
Hospitalizations | Days 15, 30, 60, and 90
  Incidence of hospitalization
Untargeted metabolomics of total plasmas and skin lesion | Days 15, 30, 60, and 90
  Changes among visits of Immune-metabolomics responses related to symptoms' incidence
Viral genomic | Day 0
  Evaluation of the pattern of viral genome of the mpox virus circulation in Brazil

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Fonseca, Study Chair — Hospital Albert Einstein
Locations (3):
- Brazil (3):
  - Hospital Universitário João de Barros Barreto, Belém, Pará
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital Naval Marcílio Dias, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No